CLINICAL TRIAL: NCT01108991
Title: Randomized Trial of Physical Activity Self-Management Intervention for Patients With COPD
Acronym: COPD-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Texas (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Coultas, Vice President for Clinical and Academic Affairs, The University of Texas Health Science Center at Tyler
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 679; R18HL092955-01A1 (NIH)
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Randomized controlled trial; Self-management support; Physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD education + Usual care (Active Comparator): Six weeks of COPD self-management education plus usual care
  Interventions: Other: COPD education + Usual care
- Physical activity self-management (Experimental): Cognitive behavioral counseling to increase lifestyle physical activity delivered over five months plus six weeks of COPD self-management education and usual care
  Interventions: Behavioral: Physical activity self-management

INTERVENTIONS:
Behavioral: Physical activity self-management — This intervention includes a manual, telephone health coach calls, and automated telephone calls. The manual has 20 chapters for the active phase and 5 maintenance phase chapters. During the first 20 weeks the health coach will call patients every other week and the automated telephone calls will occur on the alternate weeks.
  Arms: Physical activity self-management
Other: COPD education + Usual care — Six weeks of COPD self-management education plus usual care
  Arms: COPD education + Usual care

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common condition associated with major disability. There is strong evidence that pulmonary rehabilitation (PR) improves outcomes and is cost saving, but fewer than 2% of patients have access to these programs. New methods of PR are needed to increase access of patients with COPD to these established benefits. To address this gap we propose a novel physical activity self-management (PASM) program based on an evidence-based physical activity intervention designed to increase physical activity and quality of life. Key components of the program include tailored telephone counseling, a workbook, and computer-assisted telephone follow-up. We will test the following two hypotheses: 1) Patients with COPD who receive PASM have clinically and statistically significant improvements in functional performance (i.e., Chronic Respiratory Questionnaire [CRQ] dyspnea domain and 6-minute walk) compared to patients who receive UC. 2) The PASM program is more cost-effective compared to the UC. The project addresses a major gap in the current management of COPD and may provide a novel, cost-effective strategy for improving functional performance and health status.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) has been targeted nationally as a "priority" condition for which multiple strategies are needed to improve outcomes. The absolute number of years lost to disability due to COPD exceeds the years of life lost due to premature death. There is strong evidence that pulmonary rehabilitation (PR) improves outcomes and is cost saving, but fewer than 2% of patients have access to these programs. New methods of PR are needed to increase access of patients with COPD to these established benefits. To address this gap we propose a novel physical activity self-management (PASM) program based on an evidence-based physical activity intervention designed to increase physical activity and quality of life. Key components of the program include tailored telephone counseling, a workbook, and computer-assisted telephone follow-up. Our specific aims are: 1) To implement a PASM program for patients with COPD. 2) To conduct an 18-month, randomized, controlled, single-blind trial comparing PASM (n=150) to usual care (UC) (n=150) to determine the effectiveness on functional performance and health status. 3) To determine the cost-effectiveness of the intervention. Follow-up data will be collected at 6, 12, and 18 months after start of the intervention. We will test the following two hypotheses: 1) Patients with COPD who receive PASM have clinically and statistically significant improvements in functional performance (i.e., Chronic Respiratory Questionnaire [CRQ] dyspnea domain and 6-minute walk) compared to patients who receive UC. 2) The PASM program is more cost-effective compared to the UC. The project addresses a major gap in the current management of COPD and may provide a novel, cost-effective strategy for improving functional performance and health status.

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosis of COPD
* Age 45 years and older
* Affirmative response to "Are you short of breath when hurrying on the level or walking up a slight hill?"
* Post-bronchodilator FEV1/FVC <0.7 and FEV1 <70%

Exclusion Criteria:

* Inability to speak/read English
* Lives in a chronic care facility (i.e., nursing home, assisted living)
* Plans to move from the area within the next 18 months
* Life expectancy less than 12 months
* Participation in pulmonary rehabilitation or other clinical research in the past 12 months
* Inability to walk without assistance of a wheelchair or walker
* Inability to walk at least 110m on a 6-minute walk
* Uncontrolled angina, hypertension, psychiatric illness, or dementia
* Inability to obtain supplemental oxygen if indicated

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Chronic Respiratory Disease Questionnaire | 6, 12, and 18 months
  Standardized quality-of-life instrument for patients with COPD.
6-minute walk | 6, 12, and 18 months
  Standardized walking test to measure functional capacity.

SECONDARY OUTCOMES:
Cost-effectiveness | 18 months
  Health care utilization and SF-12 will be used to estimated cost effectiveness of the intervention.
Self-reported adverse event reporting | monthly for 18 months
  Patients will be asked monthly about adverse events associated with study participation.

CONTACTS AND LOCATIONS:
Overall Officials: David B Coultas, MD, Principal Investigator — VA Portland Health Care System, Oregon Health & Science University
Locations (1):
- University of Texas Health Science Center-Tyler, Tyler, Texas, United States

REFERENCES:
- [Background] Ashmore J, Russo R, Peoples J, Sloan J, Jackson BE, Bae S, Singh KP, Blair SN, Coultas D. Chronic obstructive pulmonary disease self-management activation research trial (COPD-SMART): design and methods. Contemp Clin Trials. 2013 Jul;35(2):77-86. doi: 10.1016/j.cct.2013.05.004. Epub 2013 May 13. PMID 23680985
- [Result] Jackson BE, Coultas DB, Suzuki S, Singh KP, Bae S. Rural-urban disparities in quality of life among patients with COPD. J Rural Health. 2013 Aug;29 Suppl 1(0 1):s62-9. doi: 10.1111/jrh.12005. Epub 2013 Feb 22. PMID 23944281
- [Result] Wortz K, Cade A, Menard JR, Lurie S, Lykens K, Bae S, Jackson B, Su F, Singh K, Coultas D. A qualitative study of patients' goals and expectations for self-management of COPD. Prim Care Respir J. 2012 Dec;21(4):384-91. doi: 10.4104/pcrj.2012.00070. PMID 23138844
- [Result] Russo R, Coultas D, Ashmore J, Peoples J, Sloan J, Jackson BE, Uhm M, Singh KP, Blair SN, Bae S. Chronic obstructive pulmonary disease self-management activation research trial (COPD-SMART): results of recruitment and baseline patient characteristics. Contemp Clin Trials. 2015 Mar;41:192-201. doi: 10.1016/j.cct.2015.01.018. Epub 2015 Feb 3. PMID 25657053
- [Result] Jackson BE, Coultas DB, Ashmore J, Russo R, Peoples J, Uhm M, Singh KP, Bae S. Domain-specific self-efficacy is associated with measures of functional capacity and quality of life among patients with moderate to severe chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Mar;11(3):310-5. doi: 10.1513/AnnalsATS.201308-273BC. PMID 24447029
- [Derived] Coultas DB, Jackson BE, Russo R, Peoples J, Singh KP, Sloan J, Uhm M, Ashmore JA, Blair SN, Bae S. Home-based Physical Activity Coaching, Physical Activity, and Health Care Utilization in Chronic Obstructive Pulmonary Disease. Chronic Obstructive Pulmonary Disease Self-Management Activation Research Trial Secondary Outcomes. Ann Am Thorac Soc. 2018 Apr;15(4):470-478. doi: 10.1513/AnnalsATS.201704-308OC. PMID 29283670
- [Derived] Coultas DB, Jackson BE, Russo R, Peoples J, Sloan J, Singh KP, Ashmore J, Blair SN, Uhm M, Bae S. A Lifestyle Physical Activity Intervention for Patients with Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Ann Am Thorac Soc. 2016 May;13(5):617-26. doi: 10.1513/AnnalsATS.201508-508OC. PMID 26785249